CLINICAL TRIAL: NCT03450902
Title: Combination Therapy With Chinese Herbal Formula, Yiqi Suoquan Granule, and Acupuncture for Female Mixed Urinary Incontinence
Brief Title: Chinese Herbal Therapy Combined With Acupuncture for Female Mixed Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Ran Pang, Associate Professor, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Z161100000516156
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Urinary Incontinence
Keywords: Urinary incontinence, Chinese herb, Acupuncture
MeSH Terms: conditions — Urinary Incontinence | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chinese herb & acupuncture (Experimental): Participants will take Yiqi Suoquan granule and receive acupuncture.
  Interventions: Combination Product: Chinese herb & sham acupuncture; Combination Product: Placebo & acupuncture; Other: Placebo & sham acupuncture
- Chinese herb & sham acupuncture (Active Comparator): Participants will take Yiqi Suoquan granule and receive sham acupuncture.
  Interventions: Combination Product: Chinese herb & acupuncture; Combination Product: Placebo & acupuncture; Other: Placebo & sham acupuncture
- Placebo & acupuncture (Active Comparator): Participants will take placebo granule and receive acupuncture.
  Interventions: Combination Product: Chinese herb & acupuncture; Combination Product: Chinese herb & sham acupuncture; Other: Placebo & sham acupuncture
- Placebo & sham acupuncture (Placebo Comparator): Participants will take placebo granule and receive sham acupuncture.
  Interventions: Combination Product: Chinese herb & acupuncture; Combination Product: Chinese herb & sham acupuncture; Combination Product: Placebo & acupuncture

INTERVENTIONS:
Combination Product: Chinese herb & acupuncture — Participants will take Chinese herbal formula, Yiqi Suoquan granule, which is composed of Radix Astragali 30 g, Radix Codonopsis pilosula 10g, Radix Angelica sinensis 10g, Radix Atractylodis Macrocephalae 10g, Fructus Alpiniae Oxyphyllae 10g, Radix Lindera aggregata 6g, Rhizoma Dioscoreae 10g, pericarpium citri reticulatae 10g, Rhizoma Cimicifuga 10g, Radix Bupleuri 10g, Fructus Rubi 15g, and Semen raphani 10g and prepared by the Department of Pharmacy, Guang'anmen Hospital, China Academy of Chinese Medical Sciences. Besides, Participants will receive acupuncture, three times a week. The selected acupoints include bilateral BL33, BL35, SP6, and ST36.
  Other Names: Yiqi Suoquan granule & acupuncture
  Arms: Chinese herb & sham acupuncture; Placebo & acupuncture; Placebo & sham acupuncture
Combination Product: Chinese herb & sham acupuncture — Participants will take Chinese herbal formula, Yiqi Suoquan granule, which is composed of Radix Astragali 30 g, Radix Codonopsis pilosula 10g, Radix Angelica sinensis 10g, Radix Atractylodis Macrocephalae 10g, Fructus Alpiniae Oxyphyllae 10g, Radix Lindera aggregata 6g, Rhizoma Dioscoreae 10g, pericarpium citri reticulatae 10g, Rhizoma Cimicifuga 10g, Radix Bupleuri 10g, Fructus Rubi 15g, and Semen raphani 10g and prepared by the Department of Pharmacy, Guang'anmen Hospital, China Academy of Chinese Medical Sciences. Besides, Participants will receive sham acupuncture, three times a week. The sham BL33, BL35, SP6, and ST36, which are 25 mm outward to BL33, BL35, SP6, and ST36, will be inserted with a depth of 2 to 3 mm.
  Other Names: Yiqi Suoquan granule & sham acupuncture
  Arms: Chinese herb & acupuncture; Placebo & acupuncture; Placebo & sham acupuncture
Combination Product: Placebo & acupuncture — Participants will take Chinese herbal placebo which is prepared by the Department of Pharmacy, Guang'anmen Hospital, China Academy of Chinese Medical Sciences. Besides, Participants will receive acupuncture, three times a week. The selected acupoints include bilateral BL33, BL35, SP6, and ST36.
  Other Names: placebo granule & acupuncture
  Arms: Chinese herb & acupuncture; Chinese herb & sham acupuncture; Placebo & sham acupuncture
Other: Placebo & sham acupuncture — Participants will take Chinese herbal placebo which is prepared by the Department of Pharmacy, Guang'anmen Hospital, China Academy of Chinese Medical Sciences. Besides, Participants will receive sham acupuncture, three times a week. The sham BL33, BL35, SP6, and ST36, which are 25 mm outward to BL33, BL35, SP6, and ST36, will be inserted with a depth of 2 to 3 mm.
  Other Names: placebo granule & sham acupuncture
  Arms: Chinese herb & acupuncture; Chinese herb & sham acupuncture; Placebo & acupuncture

SUMMARY:
The purpose of this study is to determine whether combination therapy with Chinese herbal formula, Yiqi Suoquan granule, and acupuncture is effective in the treatment of female mixed urinary incontinence.

DETAILED DESCRIPTION:
This factorial, randomized, controlled trial is aimed to assess the effectiveness of combination therapy with Chinese herbal formula, Yiqi Suoquan granule, and acupuncture in the treatment of female mixed urinary incontinence (MUI). Eligible participants will be randomly allocated to receiving combination therapy with Yiqi Suoquan granule and acupuncture, Yiqi Suoquan ganule plus sham acupuncture, placebo plus acupuncture, or placebo plus sham acupuncture.

To minimize the evaluation bias, the outcome assessors and statisticians will be masked to treatment allocation besides participants.

ELIGIBILITY:
Inclusion Criteria:

* (1) female, leaking with urgency and with physical activity, coughing or sneezing (MUI) for more than 1 year; (2) recorded more than 1 incontinent episode per 24 hours in their bladder diary

Exclusion Criteria:

* (1) with acute urinary tract infection; (2) with bladder outlet obstruction, (3) with neurogenic bladder (4) with interstitial cystitis, (5) with pelvic organ prolapse more than stage 2 (6) previous anti-incontinence surgery or a post-void residual urine volume more than 100 mL.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2021-04-18 (Actual); Study Completion 2021-04-18 (Actual)

PRIMARY OUTCOMES:
Change in incontinence episode per 24 h | 8 week (post-treatment) and 12 week (follow-up)
  assessed by 72 h bladder diary

SECONDARY OUTCOMES:
Change in ICIQ-SF questionnaire | 8 week (post-treatment) and 12 week (follow-up)
  assessed by ICIQ-SF questionnaire
Change in I-QOL questionnaire | 8 week (post-treatment) and 12 week (follow-up)
  assessed by I-QOL questionnaire
proportion of participants with more than 50% improvement in incontinence episodes per 24h | 8 week (post-treatment)
  assessed by 72 h bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Ran Pang, MD, Principal Investigator — Guang'anmen hospital
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The agreement for sharing IPD is not designed to be signed in informed consent form.